CLINICAL TRIAL: NCT03852966
Title: Better Sleep in Psychiatric Care - ADHD. A Pragmatic Within-group Pilot Study to Develop and Evaluate Effects and Feasibility of a CBT-based Manual for Treating Sleep Problems in Adult Patients With ADHD
Brief Title: Better Sleep in Psychiatric Care - ADHD Pilot Study
Acronym: BeSiP-ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Susanna Jernelöv, Principal Investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/2078-31/1
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Attention Deficit Disorder; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Pragmatic, within-group pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT-i/ADHD (Experimental): Behavioral treatment for sleep problems in ADHD
  Interventions: Behavioral: CBT-i/ADHD

INTERVENTIONS:
Behavioral: CBT-i/ADHD — Cognitive Behavioral Therapy for insomnia adjusted for patients with ADHD

SUMMARY:
Comorbidities, including sleep problems, are common in adult Attention Deficit Hyperactivity Disorder (ADHD). Treatment of choice for insomnia is cognitive behavioral therapy (CBT-i), but evidence is lacking for CBT-i in patients with ADHD and sleep problems.

The purpose of this study was to investigate if patients at a specialist clinic for ADHD benefit from a group delivered CBT-i treatment; whether insomnia severity improves following this treatment.

This pragmatic within-group pilot study with a pre to post and three-month follow-up design was set at a specialist psychiatric out-patient clinic for adult ADHD.

As an adjunct to care-as-usual at the clinic, a CBT-i-based group treatment targeting sleep problems prevalent in the ADHD-population, designed for patients with executive difficulties, was offered as 10 weekly 90-minute group sessions and scheduled telephone support.

All outcome measures were subjectively reported by participants. Data analyzed with dependent t-tests according to intent-to-treat.

ELIGIBILITY:
Inclusion Criteria:

* being a patient at the clinic (i.e. having a diagnosis of AD(H)D)
* self-reported sleep problems
* returning pre-treatment questionnaires and signed consent form

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Change from baseline to 10 weeks
  7-item self-reported measure of insomnia severity, 0-28 Points. Higher values represents higher severity (worse outcome)
Insomnia Severity Index (ISI) | Change from baseline to 24 weeks
  7-item self-reported measure of insomnia severity, 0-28 Points. Higher values represents higher severity (worse outcome)

SECONDARY OUTCOMES:
Adult ADHD Self-Report Scale (ASRS) | Change from baseline to 10 weeks
  18-item self-reported measure of inattention and hyperactivity symptoms. Total score 0-72. Subscale inattention/hyperactivity 0-36 points per scale. Higher scores represents more severe symptoms (worse outcome).
Adult ADHD Self-Report Scale (ASRS) | Change from baseline to 24 weeks
  18-item self-reported measure of inattention and hyperactivity symptoms. Total score 0-72. Subscale inattention/hyperactivity 0-36 points per scale. Higher scores represents more severe symptoms (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Jernelöv, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of ADHD, Northern Stockholm Psychiatry, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jernelov S, Larsson Y, Llenas M, Nasri B, Kaldo V. Effects and clinical feasibility of a behavioral treatment for sleep problems in adult attention deficit hyperactivity disorder (ADHD): a pragmatic within-group pilot evaluation. BMC Psychiatry. 2019 Jul 24;19(1):226. doi: 10.1186/s12888-019-2216-2. PMID 31340804